CLINICAL TRIAL: NCT04890431
Title: Impact of Oxygen Therapy on Fatigue in Patients With Hypermobile-type Ehlers-Danlos Syndrome: a Randomised Double-blind Placebo-controlled Study
Brief Title: Impact of Oxygen Therapy on Fatigue in Patients With Hypermobile-type Ehlers-Danlos Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OXYSED
Record Dates: First submitted 2021-05-06; First posted 2021-05-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos Syndrome | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen (Experimental)
  Interventions: Drug: Oxygen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxygen — oxygen treatment (5 L/minute for 30 minutes by nasal cannula, twice/day)
  Arms: Oxygen
Drug: Placebo — ambient air not enriched with oxygen (5 L/minute for 30 minutes by nasal cannula, twice/day)
  Arms: Placebo

SUMMARY:
The hypothesis of the OXYSED study is that the delivery of 3 months of oxygen therapy via an oxygen concentrator would reduce fatigue, pain, headaches, kinesiophobia, drug intake, dyspnea, and improve walking performance, quality of sleep and quality of life of patients with Ehlers Danlos syndrome hypermobility type (EDS / HT).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years;
* Diagnosed with EDS/HT defined by the New York critieria;
* With intense fatigue defined by an FSS ≥ 4;
* Having given free and informed written consent;
* Speaking french language;
* Being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* with progressive parenchymal pulmonary pathology (pulmonary fibrosis, post-smoking emphysema);
* having an ongoing pregnancy or breastfeeding;
* who have already received oxygen therapy for the EDS / HT indication in the last 6 months;
* having a pathology that causes fatigue, which is not compensated or treated; non-exhaustive list anemia, sleep apnea syndrome, psychiatric pathologies including severe depression, organ failure (cardiac, renal, respiratory, hepatic), endocrinopathies (hypo or hyperthyroidism, diabetes), nutritional deficiencies;
* Subject to a measure for the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
FSS (Fatigue Severity Scale) score | 7 months
FSS (Fatigue Severity Scale) score | 10 months

SECONDARY OUTCOMES:
PRISM (Pictorial Representation of Illness and Self Measure) score | 7 and 10 months
SF-36 quality of life questionnaire (Short Form Heath Survey) score | 7 and 10 months
TSK (Tampa Scale Kinesiophobia) score | 7 and 10 months
walk test results | 7 and 10 months
HIT-6 (Headache Impact Test) score | 7 and 10 months
NQ (Nijmegen questionnaire ) score | 7 and 10 months
Epworth Sleepiness score | 7 and 10 months
PSQI (Pittsburgh sleep quality index) score | 7 and 10 months
HADS (Hospital Anxiety and Depression Scale) score | 7 and 10 months
NYHA (New Year Heart Association) score | 7 and 10 months
consumption of care | 7 and 10 months
  The consumption of care is defined by the presence of at least one major criterion associated or not with the minor criterion:
  * Major criteria:
    * Variation of at least one level in the frequency of use and / or in the duration of use compared to the baseline assessment concerning the use of flexible and / or rigid orthoses,
    * Variation of at least one level of the analgesic levels used compared to the baseline assessment for pain relievers.
    * Variation of at least one level in frequency compared to the baseline assessment for physiotherapy sessions.
  * Minor criterion:
    * Variation of the total daily dose compared to the baseline assessment for painkillers.
Number of oxygen therapy sessions followed by the patient | 7 and 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris Bienvenu, Principal Investigator — Hopital Saint Joseph Marseille
Locations (3):
- France (3):
  - Hopital Raymond Poincaré, Garches
  - Clinique de la Mitterie, Lille
  - Hopital Saint Joseph, Marseille